CLINICAL TRIAL: NCT05168176
Title: Bioequivalence of Dotilavir Sodium Tablets in Healthy Subjects: A Single-center, Open, Randomized, Single-dose, Crossover Study
Brief Title: Bioequivalence of Dotilavir Sodium Tablets in Healthy Subjects in the Fasting and Fed State
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: QL-YK1-045-001
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dotilavir sodium tablet (Experimental)
  Interventions: Drug: Dotilavir sodium tablet
- Dotilavir sodium tablet(Tivicay@) (Active Comparator)
  Interventions: Drug: Dotilavir sodium tablet(Tivicay@)

INTERVENTIONS:
Drug: Dotilavir sodium tablet — The subjects randomly received single oral administration of Dotilavir sodium tablet 50mg.
  Arms: Dotilavir sodium tablet
Drug: Dotilavir sodium tablet(Tivicay@) — The subjects randomly received single oral administration of Dotilavir sodium tablet 50mg.
  Arms: Dotilavir sodium tablet(Tivicay@)

SUMMARY:
The primary purpose of this study is to evaluate the bioequivalence of two dotilavir sodium tablets in the fasting and fed state. The secondary purpose of this study is to observe the safety of the test and reference preparations. An open-label, randomized, single-dose, crossover study in healthy Chinese volunteers was performed. A single oral dose of 50 mg of two dotilavir sodium tablets was administered to 64 healthy volunteers, with 36 in the fasted group and 28 consuming a high-fat diet. The evaluated pharmacokinetic parameters, including maximum concentration (Cmax), the area under the concentration-time curve (AUC0-t and AUC0-∞) were assessed for bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects ≥18 years of age, with appropriate sex ratio
* The body mass index is in the range of 19.0-27.0 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg
* The subjects have no family planning within 3 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily

Exclusion Criteria:

* Subjects with allergic constitution.
* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.
* Blood donation, massive blood loss (#400mL) or enrolled in other clinical trials 3 months prior to screening;
* Hepatitis (including hepatitis B and C), positive screening results for AIDS or syphilis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 31 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 31days
  Evaluation of Area under the plasma concentration versus time curve (AUC0-t）
Area under the plasma concentration versus time curve (AUC0-∞) | 31days
  Evaluation of Area under the plasma concentration versus time curve (AUC0-∞)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 31days
  Collection of adverse events
Incidence of abnormal blood pressure | 31 days
  Monitor both systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No